CLINICAL TRIAL: NCT00606775
Title: Carvedilol for the Prevention of Minor Cardiac Damage and Cardiac Function in Duchenne Muscular Dystrophy
Brief Title: The Preventive Efficacy of Carvedilol on Cardiac Dysfunction in Duchenne Muscular Dystrophy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzuka Hospital (Other Government)
Collaborators: Nagoya University (Other)
Responsible Party: Takao Nishizawa, Department of Cardiology, Nagoya Universtiy Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TN1966220
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2008-02-05 (Estimated); Status verified 2007-12

CONDITIONS: Duchenne Muscular Dystrophy; Cardiomyopathies
Keywords: Adrenergic beta-Antagonists; Duchenne Muscular Dystrophy; Cardiomyopathies; Troponin I
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Cardiomyopathies | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carvedilol (Experimental)
  Interventions: Drug: Carvedilol
- Control (No Intervention)

INTERVENTIONS:
Drug: Carvedilol — 2.5-5mg/day
  Other Names: Artist, Daich-Sankyo Co.Ltd
  Arms: Carvedilol

SUMMARY:
Purpose This cardiac dysfunction in patients with Duchenne muscular dystrophy is associated with minor cardiac damage as indicated by elevation of plasma cardiac troponin I (cTnI). The purpose of this study is to investigate whether the administration of Carvedilol can suppress the minor cardiac damage and prevent deterioration of cardiac function.

DETAILED DESCRIPTION:
The life span in patients with Duchenne muscular dystrophy has been extending due to the development of artificial respiratory devices. According to that, the ratio of cardiac dysfunction as a cause of death has been increasing. This cardiac dysfunction was associated with minor cardiac damage as indicated by elevation of plasma cardiac troponin I (cTnI). Furthermore, and the detection rate of cTnI plasma as revealed to be correlated with the deterioration speed of LV dysfunction assessed by serial echocardiography measurements. Accordingly, if this minor cardiac damage is suppressed, it is postulated that the progression of cardiac dysfunction can be stopped. In the cases with ventricular arrhythmia and tachycardia, we found plasma cTnI became undetectable after administration of beta-blocker. Accordingly, we investigate whether administration of beta-blocker, carvedilol can persistently suppress the minor cardiac damage and lead to suppress the deterioration of LV function. Note that his study preventive study for preserved to moderate LV dysfunction and is not intended to the beta-blocker treatment for severe LV dysfunction. Because we assume that the mechanism of elevation of cTnI is different; spontaneous in preserved to mild LV dysfunction in patients but LV wall stress in severe LV dysfunction in patients with Duchenne muscular dystrophy.

ELIGIBILITY:
Inclusion Criteria:

Male patients with Duchenne muscular dystrophy are required to meet the following criteria:

1. Aged ８ to 45 years
2. Positive plasma cardiac troponin I (0.06ng/mL) at least 4 blood measurement in every 3 month.
3. Left ventricular ejection fraction >30% by echocardiography assessment
4. Written informed consent

Exclusion Criteria:

Patients with the following conditions will be excluded from the study:

1. Left ventricular ejection fraction <30%
2. No plasma cTnI elevation
3. beta-blocker is already administered without measurement of plasma cTnI
4. Contraindication against treatment with β blockers
5. Any other serious disease that could potentially complicate the management and follow-up protocols

Ages: 8 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The suppression of minor cardiac damage indicated as elevation of plasma cTnI | 2 years

SECONDARY OUTCOMES:
Left ventricular function deterioration assessed by echocardiography In-hospital mortality for cardiac dysfunction In-hospital mortality for any cause Overall mortality | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Takao Nishizawa, MD, PhD, Principal Investigator — Department of Cardiology, Nagoya University Graduate School of Medicine
Locations (1):
- Suzuka Hospial, Suzuka, Mie-ken, Japan

REFERENCES:
- [Background] Sato Y, Yamada T, Taniguchi R, Nagai K, Makiyama T, Okada H, Kataoka K, Ito H, Matsumori A, Sasayama S, Takatsu Y. Persistently increased serum concentrations of cardiac troponin t in patients with idiopathic dilated cardiomyopathy are predictive of adverse outcomes. Circulation. 2001 Jan 23;103(3):369-74. doi: 10.1161/01.cir.103.3.369. PMID 11157687
- [Background] Yasuma F, Konagaya M, Sakai M, Kuru S, Kawamura T. A new lease on life for patients with Duchenne muscular dystrophy in Japan. Am J Med. 2004 Sep 1;117(5):363. doi: 10.1016/j.amjmed.2004.03.028. No abstract available. PMID 15336589
- [Background] Hunsaker RH, Fulkerson PK, Barry FJ, Lewis RP, Leier CV, Unverferth DV. Cardiac function in Duchenne's muscular dystrophy. Results of 10-year follow-up study and noninvasive tests. Am J Med. 1982 Aug;73(2):235-8. doi: 10.1016/0002-9343(82)90184-x. PMID 7114081
- [Background] Jefferies JL, Eidem BW, Belmont JW, Craigen WJ, Ware SM, Fernbach SD, Neish SR, Smith EO, Towbin JA. Genetic predictors and remodeling of dilated cardiomyopathy in muscular dystrophy. Circulation. 2005 Nov 1;112(18):2799-804. doi: 10.1161/CIRCULATIONAHA.104.528281. Epub 2005 Oct 24. PMID 16246949
- [Background] Ishikawa Y, Bach JR, Minami R. Cardioprotection for Duchenne's muscular dystrophy. Am Heart J. 1999 May;137(5):895-902. doi: 10.1016/s0002-8703(99)70414-x. PMID 10220639